CLINICAL TRIAL: NCT00836303
Title: A Randomized Controlled Trial of a Multilevel Intervention to Increase Colorectal Cancer Screening Among Latino Immigrants in a Primary Care Facility
Brief Title: Trial of a Multilevel Intervention to Increase Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Francesca M. Gany/Associate Professor, New York University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: T01CD000146 (NIH)
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients of physicians randomly assigned to the control group received usual care
- Intervention Group (Experimental): This group will receive the behavioral intervention.
  Interventions: Behavioral: Colorecatal Cancer Screening Activation

INTERVENTIONS:
Behavioral: Colorecatal Cancer Screening Activation — Research assistants showed intervention patients a colorectal cancer educational video in Spanish on a portable personal digital video display device while the patients were waiting for their visit. The 11-minute video was developed by the National Alliance for Hispanic Health and was accompanied by a brochure with key information from the video {http://www.hispanichealth.org/publication/}. Intervention patients were also given a one-page reminder to hand to their physicians notifying them 1) of their patients' eligibility for colorectal cancer screening, and 2) of their patients' receipt of CRC educational material.
  Arms: Intervention Group

SUMMARY:
This study will assess the effectiveness of a culturally-responsive intervention to increase colorectal cancer (CRC) screening among Latino immigrants in a primary care clinic setting of a large municipal Hospital in New York City. propose a randomized, control trial to determine if a video-based intervention, that educates and activates the patient and the provider via the patient, will increase rates of CRC screening referrals compared to a control group.

Colorectal cancer remains one of the most prevalent cancers among the general population, as well as in the Latino population, in the United States. There are serious disparities in CRC screening rates between different races and socio-demographic populations (American Cancer Society: Colorectal Cancer Facts and Figures - Special Edition 2005). Latino immigrants are one of the populations most affected by the lack of screening, reducing their relative benefit from preventive CRC services. This study will use a modified version of an intervention developed and studied by Pignone (11), with changes made to be tailored specifically to the Latino immigrant population. The outcomes measured will include referral for CRC screening and adherence with providers' referrals. In addition, the investigators will measure screening rates for other cancer screening tests to assess if the CRC intervention displaces or facilitates other cancer screening. A sample of Latino immigrants seeking care at the primary care clinic of Bellevue Hospital will be accrued through a process of consecutive sampling until reaching the proposed sample size of 101 patients in each group (alpha 0.05 and power of 80%). To analyze the effectiveness of the intervention the investigators will use the z-test and will report the difference in proportion between the intervention and the control group with a 95% CI, adjusting for intra-class correlations and covariates. A repeated measurement analysis with logistic regression will be used to examine the effects of covariates.

ELIGIBILITY:
Inclusion Criteria:

* Adult Latino immigrants
* Men and women
* 50 years and older
* Having had at least 2 previous visits to the primary care clinic in the past 2 years

Exclusion Criteria:

* Personal or family history of colorectal cancer.
* Had fecal occult blood testing (FOBT) in the past year, or flexible sigmoidoscopy or barium enema in the past 5 years, or colonoscopy in the past 10 years.
* Lower gastrointestinal symptoms, including bleeding, pain, diarrhea and/or constipation.
* Too ill to participate
* Any cancer diagnosis other than non-melanoma skin cancer.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-12; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Completion of Colorectal cancer screening | 3 months

SECONDARY OUTCOMES:
physician recommendation for colorectal cancer screening
Patient adherence to physician recommended colorectal cancer screening test | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Francesca M Gany, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.hispanichealth.org/